CLINICAL TRIAL: NCT01017458
Title: A Randomized, Double-Blind, Placebo-Controlled, Double-Dummy, Multiple-Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic Endpoints of MK0773 in Healthy Older Men
Brief Title: Safety and Tolerability of MK0773 in Healthy Older Men (0773-004)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0773-004; 2009_693; MK-0773-004
Record Dates: First submitted 2009-11-18; First posted 2009-11-20 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Healthy
Keywords: Healthy Adults
MeSH Terms: interventions — 3-fluoro-N-(3H-imidazo(4,5-b)pyridin-2-ylmethyl)-1,4a,6a-trimethyl-2-oxo-2,4a,4b,5,6,6a,7,8,9,9a,9b,10,11,11a-tetradecahydro-1H-indeno(5,4-f)quinoline-7-carboxamide; testosterone enanthate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): MK0773 + placebo injection
  Interventions: Drug: MK0773; Drug: Comparator: placebo injection
- 2 (Active Comparator): placebo to MK0773 + testosterone injection
  Interventions: Drug: Comparator: testosterone enanthate; Drug: Comparator: placebo oral tablet
- 3 (Placebo Comparator): placebo to MK0773 + placebo injection
  Interventions: Drug: Comparator: placebo oral tablet; Drug: Comparator: placebo injection

INTERVENTIONS:
Drug: MK0773 — Three 25mg oral tablets MK0773 bid, for 12 weeks
  Arms: 1
Drug: Comparator: testosterone enanthate — intramuscular injection 200mg testosterone enanthate q14d, for 12 weeks
  Other Names: Delatestryl
  Arms: 2
Drug: Comparator: placebo oral tablet — placebo oral tablet bid, for 12 weeks
  Arms: 2; 3
Drug: Comparator: placebo injection — placebo intramuscular injection q14d, for 12 weeks
  Arms: 1; 3

SUMMARY:
This study will assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of MK0773 in healthy older men.

ELIGIBILITY:
Inclusion Criteria:

* Subject is in good general health
* Subject agrees to avoid excess alcohol and strenuous physical activity during the study
* Subject who is sexually active with partners of reproductive potential agrees to use two forms of appropriate contraception during the study

Exclusion Criteria:

* Subject has significant drug allergies
* Subject has donated blood within the last 8 weeks or has taken an investigational drug in another clinical trial within the last 4 weeks
* Subject is a regular user or past abuser of any illicit drug (including alcohol)
* Subject drinks excessive amounts of caffeinated beverages
* Subject has a history of cancer
* Subject has a history of prostate or testicular surgery

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2007-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Number of subjects with Clinical Adverse Events (CAE) | 12 weeks
Number of subjects with Serious CAEs | 12 weeks
Number of subjects with drug-related CAEs | 12 weeks
Number of subjects with serious drug-related CAEs | 12 weeks
Number of subjects that discontinued with CAEs | 12 weeks
Number of subjects with Laboratory Adverse Events (LAE) | 12 weeks
Number of subjects with drug-related LAEs | 12 weeks
Number of subjects with serious LAEs | 12 weeks
Number of subjects with serious drug-related LAEs | 12 weeks
Number of subjects that discontinued with LAEs | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC